CLINICAL TRIAL: NCT04233970
Title: Development and Evaluation of an Interactive Web-based Programme on Relapse Management for People With Multiple Sclerosis - a Randomized Controlled Trial With Mixed Methods Process Evaluation
Brief Title: Development and Evaluation of a Web-based Programme on Relapse Management for People With Multiple Sclerosis
Acronym: POWER@MS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Cologne (Other); University Medical Center Goettingen (Other); Heinrich-Heine University, Duesseldorf (Other); Gaia AG (Industry); Deutsche Multiple Sklerose Gesellschaft (DMSG), Bundesverband e.V. (Unknown); MS-Stiftung Trier (Unknown); BBK Dachverband e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: POWER@MS2
Record Dates: First submitted 2020-01-02; First posted 2020-01-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing Remitting; Relapse Management; Steroids; Autonomy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted as an investigator blinded trial and participating physicians as well as MS centres in general will not be provided with any information about group assignment. Randomization will take place only after baseline documentation. Blinding of the trial participants is pursued, but only possible to a limited extent. Furthermore, it cannot be prevented that patients discuss the intervention contents with their physician. Thus participants and neurologists might realize their group assignment. While blinding in complex educational interventions including a webinar is virtually not possible, the only strategy to increase similarity of groups is to have an active control group, which we aim for with the optimized standard care group. Furthermore, the outcome assessors are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention group will receive access to the multi-component, web-based intervention programme. The intervention programme will be developed in line with principles of patient empowerment and based on the Theory of Planned Behaviour.
  Interventions: Behavioral: web-based intervention programme
- Control group (Active Comparator): Participants randomized to the control group will receive access to the web-based control programme with optimized standard care.
  Interventions: Behavioral: web-based information material offered via the same platform (broca®) in addition to usual care

INTERVENTIONS:
Behavioral: web-based intervention programme — The intervention will be designed as an individualized, dialogue-based system that will provide PwMS coordinated, individually tailored information based on the software platform broca®. The intervention programme will consist of three sections:
  1. EBPI/decision aid (five modules plus decision aid in case of an acute relapse) provided by the broca® programme. The key element of the EBPI/decision aid is the information on glucocorticosteroids for the treatment of acute relapses.
  2. A webinar led via WebEx by a trained MS nurse with questioning/chat session (approx. 60-75min).
  3. A supervised chat room provided via the DMSG (https://www.dmsg.de/ms-connect). In addition, email reminders will be used to enhance involvement of participants.
  Arms: Intervention group
Behavioral: web-based information material offered via the same platform (broca®) in addition to usual care — Participants in the control group will have access to web-based information material offered via the same platform (broca®) in addition to usual care. The control group intervention will be based on material of the German Multiple Sclerosis Society (DMSG) on relapse management. The programme will accompany the participants over a period of 4 weeks and a reminder system with neutral e-mail reminders will be used to promote the use of the programme.
  Arms: Control group

SUMMARY:
This randomized controlled trial will evaluate a web-based relapse management programme, which is easily accessible for people with multiple sclerosis. The trial is accompanied by a mixed-methods process evaluation and a health economic evaluation.

It is expected that the programme will positively change patients' relapse management and strengthen their autonomy and participation.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory, degenerative disease of the central nervous system manifesting at first with relapses in about 85% of the cases. In Germany, intravenous mostly inpatient therapy with high-dose corticosteroids is the treatment standard of acute relapses. The treatment leads to short-term faster reduction of symptoms in about 25 of 100 treated patients (absolute risk reduction), but has no long-term benefits over placebo treatment. Also intravenous treatment is not superior to oral treatment. Therefore, informed decisions on relapse management are required. An earlier randomized controlled trial (RCT) showed that evidence-based patient information (EBPI) and education on relapse management leads to significantly more informed decisions and more relapses not treated or treated with oral steroids. POWER@MS2 builds on that evidence by transferring the content to a web-platform and making the intervention easily accessible and implementable.

The intervention will be evaluated in a pragmatic double-blind (PwMS and outcome assessors) RCT. Participants will be randomized to an interactive web-based programme (intervention group) or a web-based programme with standard information on relapse management based on the contents of the German Multiple Sclerosis Society (DMSG).

POWER@MS2 aims to demonstrate fewer glucocorticoid relapse therapies, and, in case of treated relapses, less intravenous and more orally administered therapies (primary endpoint: proportion of relapses not treated or treated with oral steroids). PwMS will be recruited via all participating centres (private neurology practices and MS outpatient departments (academic and community hospitals)) in Germany. In the federal state of Schleswig-Holstein all neurologists will be contacted. Interested and eligible PwMS will be provided with a study information sheet by the participating MS centres. Informed consent will be obtained by a physician in the MS centre. After giving their informed consent, contact data (address, email, telephone) will be forwarded to the study centre (UKE) via a secure communication platform or phone. After this, baseline data will be collected and group assignment will be performed by a block randomization procedure within the database secuTrial®. After successful randomization, PwMS will receive access (login) details to the intervention or control platform within 4-6 weeks.

Participants will be monitored for at least 12 up to 36 months (on average 24 months). Every three months, measures are recorded by a standardized phone interview executed by the coordinating study centre. Recruitment will be completed after approximately nine months. The trial will end as soon as the last participant has reached 12 months of follow-up. All participants, who have not reached 36 month of follow-up, will be called for a final phone interview.

We consider the specific risks for participating PwMS to be very low. No negative effects on the quality of life of PwMS as well as disability or other undesired events due to omitted or oral steroid administration are to be expected as previous studies showed. It is more likely that there will be positive effects for trained PwMS in terms of more autonomous decision-making and differentiated use of steroids. Participants will be educated on potentially dangerous side effects of steroid therapies and their early detection by an information sheet. To assist the physician in assessing whether oral medication is acceptable, participants will be issued a certificate with documented decision-making knowledge. As part of this study, all study participants will be contacted by phone every three months. This will also allow individual risk identification and the initiation of appropriate measures if required.

Nonetheless, it could be possible that some participants feel harassed or pressured by the intervention or the permanent contact attempts. In order to detect possible adverse events, PwMS and physicians will be asked by questionnaires throughout the study as part of the process evaluation. As relevant adverse events are unlikely, no stopping rules will be applied. Nevertheless, safety measures are applied to control for anxiety, depression and disease specific quality of life. Furthermore, standard disease monitoring parameters will be collected (e.g. relapse rate, disability status) and discussed by the steering committee. Adverse effects will be documented in the secuTrial® system. Since the programme is accessed from home, there is little organisational and time expenditure. Study participants may leave the study at any time and may withdraw consent to study participation without negative consequences. Reasons will be asked for and, if provided, recorded.

The unit of analysis for the primary endpoint is the occurrence of relapses. Eighty one relapses per group yield a power of 85% at a two-tailed significance level of 5% given proportions of 78% and 56% of orally treated or non-treated relapses in the intervention group and the control group, respectively, as observed in a previous study. It is expected that these relapse rate can be observed in a total of 170 patients with 1 to 2 years follow-up, corresponding to an annual relapse rate of 0.64. The dropout rate is expected be about 10%, as in the previous study. Therefore, 188 participants will be randomized.

Data will be obtained at different time points using paper-based (primary choice) and (if requested) web-based questionnaires. First of all, informed consent and patient-related contact data will be obtained from interested PwMS in the MS centres and a copy will be send to the study centre (UKE) by regular mail. Baseline data will be obtained by participating MS centres before randomisation. From this point in time, the study centre (UKE), will take over the handling of the participants. To secure follow-up data, study participants will be contacted by the study centre via phone within the first two weeks to secure communication lines and to perform the phone interview. Student assistants will be trained on this interaction. Trial data will be collected throughout the course of the study as well as in the last follow-up in order to examine the intervention effect on the study outcomes. However, beyond 3-monthly phone interviews, major assessments will be only at baseline and after 12 months. All study relevant data will be entered in secuTrial® and provided online. PwMS and medical staff of centres as well as the central study team (defined health researchers and study assistants) can enter data.

The preparation of the declaration of consent (including voluntariness) and the handling of all data collected within the scope of the study will be carried out in accordance with the recommendations of the Ethics Committee of the University of Lübeck and the EU General Data Protection Regulation (Datenschutz-Grundverordnung, DSGVO). Data protection concerns with regard to the intervention platform will be met by securing a protected web platform. The intervention programme as well as the control programme will be provided via a secure online platform that meets all legal requirements (SSL Encryption).

All study data will be used and evaluated pseudonymously by the members of the coordinating centre and consortium partners involved. The publication of the study results and the provision of the data in an online resource will only take place in an anonymised form. Study participants will be informed about the results of the survey through a publication of the results on the DMSG website after completion of the study.

The primary endpoint is evaluated using a generalized linear model with mixed effects and logit link function. Subject specific effects are modelled as random, whereas intervention group (IG vs. CG) and study centre are included as fixed effects in the model. The intervention effect is reported as odds ratio (OR) with 95% confidence interval (CI) and p-value testing the null hypothesis of no intervention effect (i.e. OR=1). Longitudinal assessments of quality of life and impairment are analysed by means of Gaussian linear models for repeated measures (so-called mixed model for repeated measurements (MMRM)) with intervention group (IG vs. CG), time, intervention-by-time interaction, and study centre as factors and baseline score as covariate. The error terms are assumed to follow a multivariate normal distribution with unstructured covariance. Least squares mean changes from baseline will be reported for both groups with 95% CI as well as the difference between the least squares intervention group means (IG vs. CG) with 95% CI and p-value testing the null hypothesis of no treatment effect. In subgroup and regression analyses, effects of age, gender, level of education, centre and impairment will be explored.

Reasons for study withdrawal will be reported. All PwMS will be analysed in the group they were randomized to following the intention-to-treat principle. Early study discontinuations will be treated as independent right censoring in the primary analysis. In case of substantial or differential study discontinuations the validity of the independent censoring assumption will be explored in shared random effects models of the primary endpoint and time to study discontinuation. To handle missing data in baseline variables or follow-up assessments, multiple imputation models will be applied. All details of the statistical analyses including definitions of analysis populations will be prespecified in the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* clinically isolated syndrom, suspected or diagnosed relapsing remitting MS
* at least 1 relapse in the last year and/or at least 2 relapses in the last 2 years
* access to the internet and ability to use websites

Exclusion Criteria:

* primary progressive MS
* secondary progressive MS
* acute relapse
* severe visual impairment
* severe psychiatric disorder (judged based on clinical impression)
* allergic hypersensitivity to corticosteroids
* participation in the EBSIMS training programme (the relapse management training programme was offered in Hamburg and Bad Segeberg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Assessment of change in relapse treatment (relapses not treated or treated with oral steroids). | Telephone interview at month 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 after patient inclusion and after final patient reaches month 12
  Standardized questionnaire to assess change of relapses and their treatment. The questionnaire will be applied during 3-monthly phone interviews.

SECONDARY OUTCOMES:
Annual relapse rate | Telephone interview at month 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 after patient inclusion and after final patient reaches month 12
  Standardized questionnaire to assess relapses. The questionnaire will be applied during 3-monthly phone interviews (includes relapse symptoms (worsened or newly occurred), degree of impairment due to the relapse, etc.).
Relapse Risk Knowledge | Month 3 and 12 after patient inclusion
  The standardized questionnaire RiKno 2.0 was adapted to a 10-item version to assess relapse risk knowledge.
Planned Behaviour in MS Scale (PBMS relapse) | Month 3 and 12 after patient inclusion
  The validated questionnaire PBMS was adapted to a 18-item version focussiong on steroid therapy.
Control Preference Scale relapse (CPS relapse) | Month 3 after patient inclusion
  The Control Preference Scale (CPS) was adapted CPS relapse in order to assess relapse management decision-making. As a surrogate of decision quality, preferred and realized role preference in relapse management decision-making will be assessed. The scores for preferred and realized roles are grouped into active, collaborative or passive with response options ranging from A (active role in relapse mangement decision-making), over C (shared relapse management decision-making) to E (passive role in relapse management decision-making).
Patient Activation Measure (PAM) | Baseline, month 3, 12, 24, 30, 36 after patient inclusion and after final patient reaches month 12
  Standardized assessment of patient activation development (i.e. expressed in the confidence and knowledge to take action, as well as actually taking health-related action).
Impairment in the Expanded Disability Status Scale (EDSS) | Baseline and month 12 after patient inclusion
  MS impairment measurement with a score ranging from 0.0 (normal neurological exam) to 10.0 (death due to MS).
United Kingdom Neurological Disability Scale (UNDS) | Telephone interview at Baseline, month 12, 15, 18, 21, 24, 27, 30, 33, 36 after patient inclusion and after the final patient reaches month 12
  A patient-rated scale measuring impairment based on 11 subscales (memory, mood, vision, speech and communication, swallow, use of arms, use of legs, bladder, bowel, fatigue, pain). For all subscales subscores are calculated ranging from 0 (no impairment) to 5 (significant degree of impairment).
Hamburg Quality of life in MS Scale (HAQUAMS) | Baseline and month 12 after patient inclusion
  Assessment of MS-specific quality of life based on 8 subscales (consisting of 38 individual items) and 4 additional questions. For all subscales, average subscores are calculated from the values of the respective items (ranging from 1 to 5), with high scores standing for low quality of life and low scores standing for high quality of life.
EQ-5D | Baseline, month 3, 12, 24, 30, 36 after patient inclusion and after the final patient reaches month 12
  Assessment of health-related quality of life.
Hospital Anxiety and Depression Scale (HADS) | Baseline and month 12 after patient inclusion
  Assessment of depression and anxiety based on 14 items on 2 scales (7 on the subscale "anxiety" and 7 on the subscale "depression"), ranging from 0 (low anxiety/depression level) to 3 (high anxiety/depression level) per item, resulting in a range of 0 to 21 per scale or 0 to 42 for the total HADS value.
Health Economic Evaluation | Telephone interview at Baseline, month 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 after patient inclusion and after the final patient reaches month 12
  Assessment of all direct costs associated with the intervention as well as costs resulting from the consumption of health-related goods and services as well as indirect costs due to productivity losses.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Köpke, Prof., Principal Investigator — Institute of Nursing Science, University of Cologne; Anne C Rahn, Prof., Principal Investigator — Institute of Social Medicine and Epidemiology, Nursing Research Unit, University of Lübeck
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
An anonymised data set will be published in major journals in order to disseminate the study results. In addition, all trial results will be communicated at scientific conferences and meetings (e.g. at the yearly DGN congress) by the investigators and presented on the DMSG website and other relevant patient websites.
Supporting Information: Study Protocol
URL: https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-021-05059-1

REFERENCES:
- [Background] Kopke S, Kasper J, Muhlhauser I, Nubling M, Heesen C. Patient education program to enhance decision autonomy in multiple sclerosis relapse management: a randomized-controlled trial. Mult Scler. 2009 Jan;15(1):96-104. doi: 10.1177/1352458508095921. Epub 2008 Oct 9. PMID 18845657
- [Background] Kopke S, Richter T, Kasper J, Muhlhauser I, Flachenecker P, Heesen C. Implementation of a patient education program on multiple sclerosis relapse management. Patient Educ Couns. 2012 Jan;86(1):91-7. doi: 10.1016/j.pec.2011.03.013. Epub 2011 Apr 19. PMID 21507595
- [Background] Heesen C, Kasper J, Segal J, Kopke S, Muhlhauser I. Decisional role preferences, risk knowledge and information interests in patients with multiple sclerosis. Mult Scler. 2004 Dec;10(6):643-50. doi: 10.1191/1352458504ms1112oa. PMID 15584489
- [Background] Ajzen I. The theory of planned behaviour: reactions and reflections. Psychol Health. 2011 Sep;26(9):1113-27. doi: 10.1080/08870446.2011.613995. PMID 21929476
- [Background] Kopke S, Kern S, Ziemssen T, Berghoff M, Kleiter I, Marziniak M, Paul F, Vettorazzi E, Pottgen J, Fischer K, Kasper J, Heesen C. Evidence-based patient information programme in early multiple sclerosis: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2014 Apr;85(4):411-8. doi: 10.1136/jnnp-2013-306441. Epub 2013 Oct 8. PMID 24104856
- [Background] Hawkins RP, Kreuter M, Resnicow K, Fishbein M, Dijkstra A. Understanding tailoring in communicating about health. Health Educ Res. 2008 Jun;23(3):454-66. doi: 10.1093/her/cyn004. Epub 2008 Mar 17. PMID 18349033
- [Background] Kasper J, Kopke S, Fischer K, Schaffler N, Backhus I, Solari A, Heesen C. Applying the theory of planned behaviour to multiple sclerosis patients' decisions on disease modifying therapy--questionnaire concept and validation. BMC Med Inform Decis Mak. 2012 Jul 2;12:60. doi: 10.1186/1472-6947-12-60. PMID 22747904
- [Background] Zill JM, Dwinger S, Kriston L, Rohenkohl A, Harter M, Dirmaier J. Psychometric evaluation of the German version of the Patient Activation Measure (PAM13). BMC Public Health. 2013 Oct 30;13:1027. doi: 10.1186/1471-2458-13-1027. PMID 24172020
- [Background] Stepleman L, Rutter MC, Hibbard J, Johns L, Wright D, Hughes M. Validation of the patient activation measure in a multiple sclerosis clinic sample and implications for care. Disabil Rehabil. 2010;32(19):1558-67. doi: 10.3109/09638280903567885. PMID 20590506
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Gold SM, Heesen C, Schulz H, Guder U, Monch A, Gbadamosi J, Buhmann C, Schulz KH. Disease specific quality of life instruments in multiple sclerosis: validation of the Hamburg Quality of Life Questionnaire in Multiple Sclerosis (HAQUAMS). Mult Scler. 2001 Apr;7(2):119-30. doi: 10.1177/135245850100700208. PMID 11424632
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Derived] Wenzel L, Heesen C, Peper J, Grentzenberg K, Fasshauer E, Scheiderbauer J, Thale F, Meyer B, Kopke S, Rahn AC. An interactive web-based programme on relapse management for people with multiple sclerosis (POWER@MS2) - development, feasibility, and pilot testing of a complex intervention. Front Neurol. 2022 Sep 23;13:914814. doi: 10.3389/fneur.2022.914814. eCollection 2022. PMID 36212638
- [Derived] Wenzel L, Heesen C, Scheiderbauer J, van de Loo M, Kopke S, Rahn AC. Evaluation of an interactive web-based programme on relapse management for people with multiple sclerosis (POWER@MS2): study protocol for a process evaluation accompanying a randomised controlled trial. BMJ Open. 2021 Oct 1;11(10):e046874. doi: 10.1136/bmjopen-2020-046874. PMID 34598981
- [Derived] Rahn AC, Wenzel L, Icks A, Stahmann A, Scheiderbauer J, Grentzenberg K, Vomhof M, Montalbo J, Friede T, Heesen C, Kopke S. Development and evaluation of an interactive web-based decision-making programme on relapse management for people with multiple sclerosis (POWER@MS2)-study protocol for a randomised controlled trial. Trials. 2021 Feb 14;22(1):139. doi: 10.1186/s13063-021-05059-1. PMID 33583424

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04233970/SAP_000.pdf